CLINICAL TRIAL: NCT02772354
Title: Radiofrequency Ablation of Symptomatic Frequent Ventricular Premature Complexes as a First-line Therapy in Pediatric Population Without Structural Heart Disease
Brief Title: Radiofrequency Ablation of Symptomatic Frequent Ventricular Premature Complexes in Pediatric Population
Acronym: RAS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ILM511
Record Dates: First submitted 2016-04-15; First posted 2016-05-13 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Ventricular Arrhythmia
Keywords: Pediatric population, ablation
MeSH Terms: interventions — Catheter Ablation; Metoprolol; Verapamil

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Ablation (Experimental): Standard radiosurgery ablation of premature ventricular complexes using navigation system.
  Interventions: Procedure: Radiofrequency catheter ablation; Device: NAVI-STAR® RMT ThermoCool
- Control (Active Comparator): Antiarrhythmic therapy of premature ventricular complexes according to the guidlines
  Interventions: Drug: Metoprolol; Drug: Verapamil

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation — Biosense Webster: NAVI-STAR ThermoCool, NAVI-STAR® RMT ThermoCool
  Arms: Ablation
Drug: Metoprolol — Antiarrhythmic therapy of premature ventricular complexes
  Metoprolol 12-50 mg
  Arms: Control
Drug: Verapamil — Verapamil 20-240 mg
  Arms: Control
Device: NAVI-STAR® RMT ThermoCool
  Arms: Ablation

SUMMARY:
To evaluate the effectiveness and safety of catheter ablation of frequent symptomatic PVCs in the pediatric population as first-line therapy compared with antiarrhythmic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, frequent, premature ventricular complexes (more than 10,000 according to the 24 hour Holter ECG)

Exclusion Criteria:

* Antiarrhythmic therapy before inclusion Structural heart pathology requiring surgical correction; Premature ventricular complexes associated with structural heart disease; Previously performed radiofrequency ablation due to premature ventricular complexes.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-09 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The presence of premature ventricular complexes ≥ 300 according to the 24-hour Holter ECG monitoring | 12 months

SECONDARY OUTCOMES:
Complications | 12 months
Left ventricle diameter | 12 months
Right ventricle diameter | 12 months
Premature ventricular complexes burden according to the 24- hour Holter ECG | 12 months
Ventricular tachycardia according to the 24- hour Holter ECG | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Research Clinical Institute of Pediatrics, N.I. Pirogov Russian National Research Medical University, Moscow
  - State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk